CLINICAL TRIAL: NCT06747819
Title: Effect of Cervical Epidural Steroid Injection With Neural Mobilization in Patients With Cervical Radicular Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/765
Record Dates: First submitted 2024-12-13; First posted 2024-12-24 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Cervical Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group I (Experimental)
  Interventions: Diagnostic Test: Cervical Epidural Steroid Injection (CESI)
- Interventional group II (Active Comparator)
  Interventions: Combination Product: Neural Mobilization (NM)

INTERVENTIONS:
Diagnostic Test: Cervical Epidural Steroid Injection (CESI) — Participants in this group received CESI to reduce inflammation and alleviate pain in the cervical nerve roots.
  Arms: Interventional group I
Combination Product: Neural Mobilization (NM) — Participants in this group underwent NM exercises aimed at improving nerve mobility and reducing symptoms related to nerve compression.
  Arms: Interventional group II

SUMMARY:
This study examines the effectiveness of cervical epidural steroid injections (CESI) and neural mobilization (NM), individually and in combination, in alleviating cervical radicular pain-a condition characterized by nerve root compression or irritation often due to herniated discs or bony spurs. Cervical radiculopathy leads to chronic pain, sensory and motor deficits, and disability in the upper limbs.

DETAILED DESCRIPTION:
The study is a randomized controlled trial conducted between April and October 2024, with patients diagnosed with cervical radicular pain randomized into three groups: CESI-only, NM-only, and combined CESI and NM.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18-65 years, diagnosed with chronic cervical radicular pain.
* Patients with chronic cervical radicular pain (>6 months).
* Patients who had been confirmed through clinical examination and imaging studies (MRI or CT) showed evidence of nerve root compression.
* Participants were included if they provided written informed consent, demonstrated the ability to adhere to the study protocol, and committed to attending follow-up appointments while completing the required outcome measures.

Exclusion Criteria:

* Patient refusal.
* Patients above the age of 65 were eliminated to reduce confounding by age-related health concerns and to provide a more homogenous study population for more accurate treatment outcomes.
* Patients with a history of cervical spine surgery, Uncontrolled Diabetes Mellitus, Hypertension Ischemic Heart Disease, and Pregnancy
* Patients with chronic pain syndromes that may interfere with cervical radicular pain evaluation, such as fibromyalgia, rheumatoid arthritis, or hypersensitivity, will be excluded. These disorders will be evaluated during screening using a complete medical history review, physical examination, and precise diagnostic criteria to guarantee correct detection of cervical radicular discomfort.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Numeric Pain Rating Scale (NPRS) | 12 Months
  Participants will rate their pain intensity on a scale of 0 to 10, with 0 indicating no pain and 10 indicating the worst possible pain. This measure will assess changes in pain levels from baseline through various follow-up points.
The Neck Disability Index (NDI) | 12 months
  The NDI consists of ten questions in the following domains: Pain Intensity, Personal Care, Lifting, Reading, Headaches, Concentration, Work, Driving, Sleeping, and Recreation.
  Each question contains six answer choices, scored from 0 (no disability) to 5 (complete disability

CONTACTS AND LOCATIONS:
Locations (1):
- Ghurki trust and teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No